CLINICAL TRIAL: NCT03107481
Title: Acetaminophen 1g IV vs Hydromorphone 1mg IV for the Treatment of Acute Pain in the Emergency Department
Brief Title: Acetaminophen IV vs Hydromorphone IV in the ED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Douglas P. Barnaby, MD, MS, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-7296
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Pain, Acute
Keywords: Acetaminophen; Hydromorphone; Emergency Department; Narcotics; Analgesics, Opioid; Analgesics, Non-Narcotic
MeSH Terms: conditions — Acute Pain; Emergencies | interventions — Acetaminophen; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acetaminophen (Active Comparator)
  Interventions: Drug: Acetaminophen
- Hydromorphone (Active Comparator)
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1g IV
  Arms: Acetaminophen
Drug: Hydromorphone — Hydromorphone 1mg IV
  Arms: Hydromorphone

SUMMARY:
The purpose of the current study is to compare the analgesic efficacy of intravenous acetaminophen and intravenous hydromorphone in the treatment of acute pain in the ED.

DETAILED DESCRIPTION:
This is a randomized, double-blind placebo-controlled clinical trial comparing intravenous acetaminophen and intravenous hydromorphone in the treatment of acute pain in the Emergency Department. Enrolled subjects presenting to the ED with acute pain will be randomized to receive either acetaminophen 1g IV or hydromorphone 1mg IV.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 through 64 years of age: This is a study of adult ED patients.
* Pain with onset within 7 days: Pain within seven days is the definition of acute pain that has been used in the ED literature.
* ED attending physician's judgment that the patient's pain warrants IV opioids.
* ED attending physician's judgment that the patient has capacity to provide informed consent.
* Patients must be able to understand English or Spanish.

Exclusion Criteria:

* Use of opioids or tramadol within past 24 hours.
* Use of acetaminophen or non-steroidal anti-inflammatory medication within the previous 8 hours.
* Prior adverse reaction to opioids or acetaminophen.
* Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months results in modulation of pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, and peripheral neuropathies.
* Medical condition that might affect metabolism or opioid analgesics or acetaminophen such as hepatitis, renal insufficiency or failure, hypo- or hyper-thyroidism, Addison's or Cushing's disease
* Pregnant or breastfeeding
* Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician may alter pain perception.
* SBP <100 mmHg: Opioids can produce peripheral vasodilation that may result in orthostatic hypotension.
* HR < 60/min: Opioids can cause bradycardia.
* Oxygen saturation < 95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.
* Use of MAO inhibitors in past 30 days: MAO inhibitors have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.
* Patients using transdermal pain patches: pain patches may influence both the amount of pain patients report as well as the level of relief they obtain from other treatments.
* Taking any medication that might interact with one of the study medications, such as SSRI or tricyclic anti-depressants, antipsychotics, anti-malarial medications (quinidine or halofantrine), amiodarone or dronedarone, diphenhydramine, celecoxib, ranitidine, cimetidine, ritanovir, terbinafine or St. John's Wort.
* Patients who have been previously enrolled in this same study: Patients may only be enrolled once.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2017-06-04 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
NRS Change at 60 minutes | 60 minutes
  Between group difference in change in NRS pain scores from baseline

SECONDARY OUTCOMES:
Forego Additional Pain Medication | 60 minutes
  Difference in proportion of patients who choose to forego additional pain medication
Receive Rescue Medication | Before 60 minutes
  Difference in proportion of patients who receive additional pain medication before primary outcome
Experience Medication Side Effects | 120 Minutes
  Difference in proportion of patients who experience medication side effects grouped by GI (vomiting, nausea), dermatologic (pruritis, rash), and CNS (dizziness, drowsiness) categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barnaby DP, Chertoff AE, Restivo AJ, Campbell CM, Pearlman S, White D, Bijur PE, Gallagher EJ. Randomized Controlled Trial of Intravenous Acetaminophen Versus Intravenous Hydromorphone for the Treatment of Acute Pain in the Emergency Department. Ann Emerg Med. 2019 Feb;73(2):133-140. doi: 10.1016/j.annemergmed.2018.06.019. Epub 2018 Aug 14. PMID 30119941